CLINICAL TRIAL: NCT01110486
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABT-348 as Monotherapy, in Combination With Carboplatin or in Combination With Docetaxel in Subjects With Advanced Solid Tumors
Brief Title: ABT-348 as Monotherapy or Combination With Carboplatin or Docetaxel to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-944
Record Dates: First submitted 2010-03-26; First posted 2010-04-26 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — ilorasertib; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Monotherapy, once daily (Experimental)
  Interventions: Drug: ABT-348
- Combination with carboplatin (Experimental)
  Interventions: Drug: ABT-348 and carboplatin
- Combination with docetaxel (Experimental)
  Interventions: Drug: ABT-348 and docetaxel
- Monotherapy, twice daily (Experimental)
  Interventions: Drug: ABT-348
- IV Monotherapy, once daily (Experimental)
  Interventions: Drug: ABT-348

INTERVENTIONS:
Drug: ABT-348 — An oral dose of ABT-348, once daily on Day 1, Day 8, and Day 15 of each 28 day cycle.
  Arms: Monotherapy, once daily
Drug: ABT-348 and carboplatin — An oral dose of ABT-348 will begin in Cycle 2on Day 1 and Day 8; and an IV dose of carboplatin (AUC 5.0) on Day 1 of each 21-day cycle.
  Arms: Combination with carboplatin
Drug: ABT-348 and docetaxel — ABT-348 dosing will begin in Cycle 2. An oral dose of ABT-348 on Day 1 and Day 8; and an IV dose of docetaxel (75 mg/m2) on Day 1 of each 21-day cycle.
  Arms: Combination with docetaxel
Drug: ABT-348 — An oral dose of ABT-348, twice daily on Day 1, Day 8, and Day 15 of each 28 day cycle
  Arms: Monotherapy, twice daily
Drug: ABT-348 — An IV administration of ABT-348 two hour infusion on Day 1, Day 8 and Day 15 of each 28 day cycle.
  Arms: IV Monotherapy, once daily

SUMMARY:
The purpose of this study is to determine the safety, pharmacokinetics and maximum tolerated dose of ABT-348 as monotherapy and when given in combination with carboplatin or docetaxel.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the safety, pharmacokinetics and maximum tolerated dose of ABT-348 as monotherapy and when given in combination with carboplatin or docetaxel. The secondary purpose of this study is to evaluate safety at the recommended Phase 2 dose and evaluate preliminary efficacy data regarding objective response rate time to progression, duration of overall response, and ECOG performance status of ABT-348 as monotherapy and when given in combination with carboplatin or docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of locally advanced or metastatic solid tumor.

   * That is either refractory after standard of care therapy for the disease for which standard of care therapy is not reliably effective or does not exists, or
   * For which carboplatin has been determined to be an appropriate therapy, per the investigator, or
   * For which docetaxel has been determined to be an appropriate therapy, per the investigator.
2. Eastern Cooperative Oncology Group Status of 0-2
3. Serum creatinine value of ≤ 1.5 times the upper limit of normal (ULN) and either an estimated creatinine clearance value as determined by the Cockcroft-Gault formula or based on a 24 hour urine collection creatinine clearance value of ≥ 50 mL/min
4. Adequate liver function as demonstrated by serum bilirubin < 2 x ULN and AST and ALT ≤ 2.5 x ULN
5. Adequate bone marrow as demonstrated by absolute neutrophil count (ANC) ≥ 1,500/mm2 (1.5 x 109/L); Platelets ≥ 100,000/mm2 (100 x 109/L); Hemoglobin ≥ 9.0 g/dL (1.4 mmol/L)
6. QTc interval < 500 msec
7. Left Ventricular Ejection Fraction > 50%
8. Women of child-bearing potential and men must agree to use adequate contraception (one of the following listed below) prior to the study entry, for the duration of study participation and up to 3 months following completion of therapy.
9. Capable of understanding and complying with parameters as outlined in the protocol and able to sign informed consent, approved by an Institutional Review Board (IRB) prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Subject has known active CNS involvement. The subject has untreated brain or meningeal metastases.
2. Subject has received anti-cancer therapy within a period of 21 days or 5 half lives (whichever is shorter) prior to Study Day 1
3. Subject has unresolved toxicities from prior anti-cancer therapy, grade 2 or higher clinically significant toxicity (excluding alopecia)
4. Subject has had major surgery within 28 days prior to Study Day 1
5. Subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure > 90 mmHg or systolic blood pressure > 140 mmHg
6. Subject has proteinuria grade > 1 7. Subject is receiving therapeutic anticoagulation therapy. Low dose anti coagulation (e.g., low dose heparin or warfarin) for catheter prophylaxis will be permitted.

8. Clinically significant uncontrolled condition(s) 9.Psychiatric illness/social situation that would limit compliance with study requirements 10. Subject has a known infection with HIV, Hepatitis B or Hepatitis C 11. Subject with poorly controlled diabetes mellitus 12. Subject enrolled in Arm A, B, C and D is unable to swallow or absorb oral tablets normally 13. Any medical condition which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities 14. Female subjects who are lactating or pregnant 15. Subject enrolled in Arm E has hypersensitivity to drugs formulated with polyethoxylated castor oli (Cremophor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determine the safety profile (Adverse events by toxicity grade and relationship to study drug, serious adverse events, adverse events leading to discontinuation and relevant clinical laboratory abnormalities) of ABT-348 as monotherapy or in combination | At each treatment visit
Study the pharmacokinetic of ABT-348 | At study visits
Dose limiting toxicity determination | At each treatment visit until dose-limiting toxicities observed

SECONDARY OUTCOMES:
Evaluate safety at the recommended Phase 2 dose (RPTD) and schedule of ABT-348 as monotherapy, when in combination with carboplatin or in combination with docetaxel. | At RPTD treatment visit
Evaluate preliminary efficacy data regarding objective response rate (ORR), time to progression (TTP), duration of overall response, and ECOG performance status of ABT-348 as monotherapy, when in combination with carboplatin or docetaxel. | At each treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gordon, MD, Study Director — AbbVie
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 26525, Chicago, Illinois
  - Site Reference ID/Investigator# 26524, Houston, Texas

REFERENCES:
- [Derived] Maitland ML, Piha-Paul S, Falchook G, Kurzrock R, Nguyen L, Janisch L, Karovic S, McKee M, Hoening E, Wong S, Munasinghe W, Palma J, Donawho C, Lian GK, Ansell P, Ratain MJ, Hong D. Clinical pharmacodynamic/exposure characterisation of the multikinase inhibitor ilorasertib (ABT-348) in a phase 1 dose-escalation trial. Br J Cancer. 2018 Apr;118(8):1042-1050. doi: 10.1038/s41416-018-0020-2. Epub 2018 Mar 19. PMID 29551775